CLINICAL TRIAL: NCT03625765
Title: Evaluation of an Integrated Imaging System (SmartGoggles) for in Vivo Visualization of Free Flap Perfusion Using Indocyanine Green Fluorescent Dye
Brief Title: Integrated Imaging System for In Vivo Visualization of Free Flap Perfusion Using Indocyanine Dye
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's request
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2118
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Breast Reconstruction
Keywords: Indocyanine green; SmartGoggles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SmartGoggles (Experimental): The prototype system offers real time stereoscopic fluorescence imaging along with in vivo handheld microscopy. Investigators have found that the system can detect fluorescent targets with as low as 1.2 picomoles ICG (60 nanomolar (nM) concentration). The hand-held microscopy module has a resolution of 25 micron. The prototype system has 2 complementary metal-oxide-semiconductor (CMOS) imaging sensors housed on a printed circuit board (PCB) with imaging lenses and emission filters optimized for ICG dye. The light source provides concurrent excitation centered at 780 nm and white light illumination with optical density (OD) 6 level cut-off. The SmartGoggles is a non-invasive imaging system that does not require contact with patients.
  Interventions: Device: SmartGoggles

INTERVENTIONS:
Device: SmartGoggles — the system is wearable and simulates natural binocular human vision, which minimizes the training curve for new users. The wide-field stereoscopic imaging allows clinicians to rapidly determine the extent of lesions and the hand-held microscopy probe assist clinician to visualize the lesions with high resolution.

SUMMARY:
The purpose of this study is to determine if the integrated imaging goggle (Smart Goggles) is as good as or better than current technology used to assess tissue perfusion (the extent of blood flow to the tissue) in certain types of breast reconstruction procedures.

The participants will be asked to participate in the study if they are scheduled to have a breast reconstruction procedure using a technique that involves transferring abdominal skin and tissues to the affected side of the chest. This technique is known as a breast reconstruction with a Deep Inferior Epigastric Artery Perforator (DIEP) flap.

In this pilot study, the investigators are testing the feasibility of a new device, the Integrated Imaging Goggle system (also called "Smart Goggles") as a surgical aid to differentiate between tissue with adequate blood flow and tissue without adequate blood flow by comparing measurements of fluorescence in blood vessels with current technology, the SPY-Elite system. In this study, researchers will test how quickly and accurately the fluorescent dye used to identify adequate blood flow is detected by Smart Goggles compared to the SPY Elite system.

DETAILED DESCRIPTION:
The objective is to demonstrate the sensitivity of the SmartGoggles for detection of Indocyanine (ICG) fluorescence within fasciocutaneous flap. The investigators will characterize the sensitivity of the SmartGoggles device relative to a previously validated device (the SPY Elite system).

The investigator's primary endpoint will compare the ICG transit time (the time needed for ICG to first appear in flap after intravenous injection) detected by the SmartGoggles and the SPY Elite system.

As a secondary endpoint, the investigators will compare the ICG accumulation curve and fluorescence intensity generated from each device, measured on the same region of interests (ROI). Finally, the study team will compare perfusion margin characteristics (the area between regions of well-perfused and hypoperfused tissue) as assessed by the Goggles and the SPY Elite system.

Study Design This is an unpowered pilot study to determine the sensitivity of the new SmartGoggles device for detection of ICG fluorescence in free flaps in a clinical setting. The investigators have chosen to examine ICG as the contrast agent because this agent is FDA-approved and is regularly used for evaluation of tissue perfusion. The team has chosen to use DIEP free flaps as the clinical target because these flaps are relatively large and will provide adequate surface area for measurement of fluorescent margins and comparison of fluorescence between the Goggles and SPY Elite systems.

This study will enroll 25 patients. After signing consent form all patients will undergo standard of care preoperative and postoperative evaluations. Investigators will perform one ICG angiography per patient: intraoperatively after designing and harvesting the flap. All measurements will be taken by SmartGoggles and SPY Elite systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral DIEP flap breast reconstruction
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant women
* Patients with severe hepatic insufficiency
* Patients with a history of allergic reactions or know hypersensitivity to ICG and iodide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ICG transit time detected by the SmartGoggles and the SPY Elite system. | At the end of surgery - 1 day
  The time needed for ICG to first appear in flap after intravenous injection

SECONDARY OUTCOMES:
Difference in the ICG accumulation curve and fluorescence intensity generated from each device, measured on the same region of interests | At the end of surgery - 1 day
  compared between SmartGoggles and the SPY Elite System using a one-sided non-inferiority analysis based on a paired t-test.
Difference in square area of perfusion as detected by ICG angiography under the SmartGoggles and SPY Elite systems | At the end of surgery - 1 day
  This perfusion margin characteristic provides a difference in detection by the two imaging systems

CONTACTS AND LOCATIONS:
Overall Officials: Risal Djohan, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States